CLINICAL TRIAL: NCT04574804
Title: Effects of an Online Training Program for Physiotherapists About Weight Management for People With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Kim Bennell, Prof. Kim Bennell, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UMelbourne
Record Dates: First submitted 2020-09-22; First posted 2020-10-05 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis; Overweight and Obesity
MeSH Terms: conditions — Osteoarthritis; Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomisation of participants will be conducted by a researcher with no direct involvement in the study. The biostatistician will analyse blinded, de-identified data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online training program (Experimental): online training program Participants receive access to online training program consisting of 6 e-learning modules on topics of weight management in osteoarthritis, which they will be instructed to and encourage to complete over the 6 intervention period.
  Interventions: Other: Online training program in weight management for osteoarthritis
- control group (No Intervention): control group Participants do NOT receive access to the online training program consisting of 6 e-learning modules on topics of weight management in osteoarthritis during the intervention period.

INTERVENTIONS:
Other: Online training program in weight management for osteoarthritis — An evidence based online education training program for physiotherapists in weight management for osteoarthritis. Training modules cover the following topic areas:
  1. Overweight and obesity and osteoarthritis
  2. Overview of weight regulation, overweight and obesity
  3. Examining weight stigma in physiotherapy and personal beliefs about weight
  4. Communication approach for addressing weight management
  5. Interventions for weight management
  6. Health behaviour change support
  These 6 e-learning modules comprise the online training program, access to which comprises the study intervention.
  Arms: online training program

SUMMARY:
A randomized controlled trial for which the primary objective is to evaluate the effects of an online training program on physiotherapist's self-reported confidence in knowledge about weight management for people with osteoarthritis. 80 physiotherapists will be recruited into the study and randomized to one of two arms a) online training program (access to training program for 6 weeks) or b) control group (no access to online training program during the study). Questionnaires will be completed by all participants at baseline, and again at the end of the 6 week intervention period. A biostatistician will analyse blinded, de-identified data.

DETAILED DESCRIPTION:
The Centre for Health Exercise and Sports Medicine at the University of Melbourne have developed a 6-module online training program designed to up-skill physiotherapists in weight management for osteoarthritis patients. This is a randomised controlled trial evaluating the effectiveness of the training program on physiotherapist's confidence in weight management for osteoarthritis patients. After providing informed consent and baseline data, physiotherapists will be randomized to either a) an online training program or b) control group. Those randomized to the online training group will be provided access to the a 6-module weight management training program and have six weeks to complete all the modules. Those randomized to the control group will receive no intervention. At baseline and six weeks, primary and secondary outcome measures will be completed in both groups.

The research question is: What are the effects of an online training program designed to up-skill physiotherapists in weight management for people with osteoarthritis? The primary objective is to evaluate the effects of an online training program on physiotherapist's self-reported confidence in knowledge about weight management for people with osteoarthritis.

80 participants will be recruited and randomization into the two study groups. To detect an effect size of 0.8 with 80% power and two sided significance level of 5%, 26 participants are required per group. Assuming a 35% loss to follow up, this will increase the same size to 40 per group (80 in total). The study will be conducted through The University of Melbourne. Participants will be able to access the training remotely in their own time and access all outcome measures online.

A biostatistician will analyse blinded, de-identified data. Analyses will be conducted with participants in assigned groups, with multiple imputation to account for missing data if required. Changes in self-reported confidence scores (primary outcome) will be compared between groups at 6 weeks using linear regression (with group as a factor) adjusting for baseline scores and the stratifying variables. Similar analyses will be conducted for secondary outcomes measured at baseline and 6 weeks. Process measures will be described in terms of mean (SD)/median (IQ range) or number (frequency). Standard diagnostic plots will be used to verify model assumptions.

If an imbalance is noted between groups for relevant baseline characteristics, sensitivity analyses will be conducted including these characteristics as covariates in the models assessing treatment effects.

The biostatistician will also conduct planned exploratory analyses to investigate potential moderators that could influence the effect of the training at 6 weeks. Pre-identified potential moderators include practice location (predominantly private vs predominantly public), baseline self rated confidence in weight management and years of clinical experience. To assess the moderation of the effect of randomised treatment group by the binary potential moderator (practice location), an interaction term between randomised group and the potential moderator, as well as terms for the randomised group and the potential moderator, will be included in the outcome regression model. To assess the moderation of the effect of randomised treatment group by continuous potential moderators (self rated confidence in weight management and years of clinical experience), the multivariable fractional polynomial interaction approach will be applied. This approach allows for nonlinear functional forms of the continuous potential moderator to be included in the regression model for outcomes, with the potential for separate nonlinear functional forms in each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Currently registered with the Australian Health Practitioner Registry
* Have access to a computer with internet connection
* Willing to commit to completion of an 8-10 hour online training module if randomized to the intervention group
* Willing to refrain from participating in any weight management professional development activity external to the study for six weeks of intervention
* Able to give informed consent and to commit and participate fully in the assessment and evaluation procedures over the six week period.

Exclusion Criteria:

* n/a

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Self-reported confidence in knowledge about weight management for patients with osteoarthritis | Change from baseline at 6 weeks post randomization
  Measured using an expert-developed, customized self-reported questionnaire exploring physiotherapists' perceived confidence in knowledge about weight management in osteoarthritis. Total score out of 70 possible points calculated from the responses to 14 Likert Scale (1-5) questions where higher values indicate higher confidence and lower values lower confidence in knowledge

SECONDARY OUTCOMES:
Self-reported confidence in clinical skills for weight management for patients with osteoarthritis | Change from baseline at 6 weeks post randomization
  Measured using an expert-developed, customized self-reported questionnaire exploring physiotherapists' perceived confidence in clinical skills for weight management in osteoarthritis. Total score out of 45 possible points calculated from the responses to 9 Likert Scale (1-5) questions where higher values indicate higher confidence and lower values lower confidence in clinical skills.
Self-perceived competence in nutrition care to patients with chronic disease | Change from baseline at 6 weeks post randomization
  Measured using the NUTCOMP Questionnaire, a validated six section questionnaire (four sections scored, two unscored) developed to explore health care professional's perceived competence of the provision of nutrition care. Total score out of 175 possible points calculated from the responses to the Likert Scale (1-5) for each of the 35 questions, where higher values indicate higher confidence and lower values, lower confidence.
Weight stigmatized attitudes | Change from baseline at 6 weeks post randomization
  Measured by the Anti-Fat Attitudes questionnaire which comprises 13 statements about beliefs about weight (categorized under Dislike, Fear and Willpower) which respondents answer on a 10 point 0-9 Likert type scale, where 0 = very strongly disagree and 9 = very strongly agree. Total score calculated by response to each statement out of eight. The 3 subscales (dislike, fear and willpower) will also be reported.

OTHER OUTCOMES:
Completion of training modules (process measure) | Throughout 6 week intervention period
  Data will be collected through the learning management system platform. Completion of module will be categorized by passing end of module quiz with 100%. (Repeat attempts allowed). Number of modules completed reported.
Usefulness of modules (process measure) | Throughout 6 week intervention period
  Self-reported using bespoke 4-item questionnaire upon completion of each module. Measured using a 5-point Likert scale from 1= strongly disagree to 5 = strongly agree. Items scored individually, higher scores for each item represent positive impressions towards training
Structure and content of modules (process measure) | Throughout 6 week intervention period
  Impressions of module length and module content self reported using two custom questions, each assessed as one of 3 multi-choice options. Results for each multichoice option presented as a percentage for the 2 custom questions
Time to complete each module (process measure) | Throughout 6 week intervention period
  Self-reported upon completion of each individual module (built into module quiz). Reported in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kim Bennell, PhD, BAppSci, Principal Investigator — University of Melbourne
Locations (1):
- University of Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Derived] Allison K, Jones S, Hinman RS, Briggs AM, Sumithran P, Quicke J, Holden M, Chiavaroli N, Crofts S, George E, Foster N, Bennell K. Effects of an Online Education Program on Physical Therapists' Confidence in Weight Management for People With Osteoarthritis: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2023 Apr;75(4):835-847. doi: 10.1002/acr.24828. Epub 2022 Dec 12. PMID 34931477